CLINICAL TRIAL: NCT04883047
Title: Evaluation of the Effects of Practices Performed in Accordance With the Algorithm of Coping With Birth Pain on Coping With Birth Pain, Birth Satisfaction and Birth Fear: A Randomized Controlled Study
Brief Title: The Effectiveness of the Applications Made in Line With the Algorithm for Coping With Labor Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Pinar Akbas, Expert Nurse, Doctoral student, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: laborpain
Record Dates: First submitted 2021-04-26; First posted 2021-05-12 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Labor Pain
Keywords: coping with labor pain; birth satisfaction; fear of birth
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Intervention Model Description: The study was planned as a single center stratified block parallel group randomized controlled experimental study.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experiment (Experimental): Women in the experimental group will be given care at the first stage of labor (will start in the latent phase) using Integrated Birth Support Strategies created in line with the Algorithm for Coping with Birth Pain.
  Among the interventions made into a checklist, the interventions applied to the woman will be marked by the midwives and nurses working in the delivery room. The Scale for Coping with Birth Pain (DABS), which will be applied once in each phase (latent phase, active phase and transition phase), will guide the delivery of care; Care practices will differ depending on the woman's ability to cope with labor pain.At least 3 of each sub-heading of the physical comfort parameter, at least 1 of each sub-heading of the parameter of providing emotional comfort, at least 2 of each sub-heading of informative support and advocacy sub-parameters will be applied to pregnant women by midwives / nurses working in the delivery room.
  Interventions: Other: holistic birth support strategies
- control (No Intervention): Pregnant women assigned to the control group will be followed up with the routine care applied in the delivery room.

INTERVENTIONS:
Other: holistic birth support strategies — Holistic Birth Support Strategies are composed of birth-supporting practices that were created by Horn and D'Angelo (2017) within the scope of the "Algorithm for Coping with Birth Pain" and recommended for coping with labor pain. Holistic Birth Support Strategies; It includes four parameters: physical comfort, emotional comfort, informative support and advocacy.
  Arms: experiment

SUMMARY:
Although labor pain is a physiological and natural process, when the woman cannot cope with labor pain, the health of the mother and fetus is negatively affected. These negative effects mostly focus on the respiratory system, cardiovascular system, neuroendocrine and limbic system. During birth, the mother becomes exhausted due to pain and has to use all her energy to cope with the pain.When the mother can effectively cope with the pain of labor, she starts motherhood with a positive experience, experiences the happiness of actively participating in the birth of the baby, can participate in practices with health professionals, and the problems that can be seen in the newborn are reduced because there is no need for medication. In this respect, it is extremely important for the mother, baby and family to end the birth process in the best possible way. For this reason, nursing care includes emotional, physical, spiritual and psychosocial continuous birth support and coping with the pain of labor. In this direction, the "algorithm for coping with labor pain" developed includes the interventions that should be done to cope with the pain in labor.

DETAILED DESCRIPTION:
Pain is defined as an unpleasant emotional sensation originating from a certain part of the body, often related to tissue damage, and related to the past experiences of the person. Labor pain is an experience that is a part of a natural process, takes place in a limited time, and is perceived and experienced differently by every woman. Physiological changes during labor such as maternal age, parity, weight of mother and baby, position of the fetus, anatomical structure of the pelvis, cervical dilatation and uterine contractions; psychological factors such as perception of threats to the body or soul, culture, ethnicity, anxiety, loneliness, loss of control, fear that a painful or painful event will occur, anxiety that the baby or himself may be harmed, previous pain experiences and healthcare professionals' communication with the pregnant woman Environmental factors such as noise, lighting, and birth pain significantly affect the pregnant woman's coping with labor pain.

Although labor pain is a physiological and natural process, when the woman cannot cope with labor pain, the health of the mother and fetus is adversely affected. These negative effects mostly focus on the respiratory system, cardiovascular system, neuroendocrine and limbic system. During birth, the mother becomes exhausted due to pain and has to use all her energy to cope with the pain. When the mother cannot cope, she becomes tired, and her oxygen requirement, blood pressure and cardiac out-put increase. Fear and anxiety caused by labor pain increase the release of stress hormones such as adrenaline, noradrenaline and corticosteroid. These hormones reduce the blood flow to the uterus and cause distress in the fetus by reducing the amount of oxygen in the placental flow. In addition, due to the increased adrenaline, it causes a decrease in the amount of oxytocin during delivery. This causes prolongation of labor and more bleeding. At the same time, when the woman is able to cope with labor pain, the formation of tetany in the pregnant woman is prevented by preventing hyper ventilation and hypocapnia formation.

When the mother can effectively cope with the pain of labor, she starts motherhood with a positive experience, experiences the happiness of actively participating in the birth of the baby, can participate in practices with health professionals, and the problems that may be seen in the newborn are reduced since there is no need for medication. In this respect, it is extremely important for the mother, baby and family to end the birth process in the best possible way. For this reason, nursing care includes emotional, physical, spiritual and psychosocial continuous birth support and coping with the pain of labor. Providing non-pharmacological pain relief methods such as relaxation and breathing exercises, massage, positioning, therapeutic communication, listening to music, hot-cold application, partner and family support, providing home environment is associated with a positive birth experience. Accordingly, the "algorithm for coping with labor pain" developed by Roberts et al. (2010) includes the interventions that should be done to cope with the pain at birth. The algorithm for coping with labor pain has two branches. One is the arm that shows pregnant ways of coping with pain, such as rhythmic activity, deep breathing, inner focus, relaxation between contractions, which gives clues to healthcare professionals; Another is the arm that enables the evaluation of the findings that show that the woman cannot cope with labor pain such as clenching her teeth, crying, and inability to focus. According to the algorithm, when a woman can cope with labor pain, there is no need to do any intervention. However, when the woman cannot cope with labor pain, it is easier for the woman to cope with labor pain with holistic birth support strategies such as providing physical comfort, emotional comfort, informative support and advocacy.

ELIGIBILITY:
Inclusion Criteria:

* Being in the latent phase of labor
* Not being a risky pregnant (gestational diabetes, hypertension, preeclampsia etc.)
* Not having any communication problems (mental, auditory, visual, etc.)

Exclusion Criteria:

* Pregnancy does not do the post-test applications
* Not wanting to participate in interventions applied in line with the algorithm for coping with labor pain
* Willing to leave the research
* Delivery by cesarean section

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-06-25 (Actual)

PRIMARY OUTCOMES:
Birth satisfaction as assessed by the Birth Satisfaction Scale | will be measured in the first 6 hours postpartum
  Measurements will be made using the Birth Satisfaction Scale.The total number of points to be obtained from the scale varies between 30 and 150 points, but the scale does not have a cut-off point. As the scores obtained from the scale increase, the level of birth satisfaction increases.
Fear of childbirth as assessed by the Wijma Birth Expectation/Experience Scale-Version B | will be measured in the first 6 hours postpartum
  Measurements will be made using the Wijma Birth Expectancy / Experience Scale Version B. While the minimum score on the scale is 33, the maximum score is 198. The high scores indicate that the fear of childbirth experienced by women is high.

CONTACTS AND LOCATIONS:
Overall Officials: Şengül YAMAN SÖZBİR, PhD, Principal Investigator — Gazi Universty
Locations (1):
- Karabük Training and Research Hospital, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR